CLINICAL TRIAL: NCT00006350
Title: Allogeneic Hematopoietic Stem Cell Transplantation for Hematologic Malignancies After a Non-Myeloablative Conditioning Regimen From HLA-Matched Sibling Donors
Brief Title: Mycophenolate Mofetil, Tacrolimus, Daclizumab, and Donor Peripheral Stem Cell Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: MSGCC-0012; CDR0000068212 (Registry Identifier: PDQ (Physician Data Query)); NCI-V00-1624
Record Dates: First submitted 2000-10-04; First posted 2004-03-08 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: recurrent adult Hodgkin lymphoma; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; recurrent mantle cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Daclizumab; Mycophenolic Acid; Tacrolimus; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: daclizumab
Biological: therapeutic allogeneic lymphocytes
Drug: mycophenolate mofetil
Drug: tacrolimus
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Monoclonal antibodies such as daclizumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Peripheral stem cell transplantation from a brother or sister may be effective treatment for hematologic cancer. Sometimes the transplanted cells can be rejected by the body's tissue. Mycophenolate mofetil, tacrolimus, and donor white blood cells may prevent this from happening.

PURPOSE: Phase II trial to study the effectiveness of mycophenolate mofetil, tacrolimus, daclizumab, and donor peripheral stem cell transplantation in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether donor hematopoiesis can be safely established using a nonmyeloablative conditioning regimen followed by HLA matched sibling donor peripheral blood stem cell transplantation in patients with hematologic malignancies. II. Determine whether mixed chimerism can be safely converted to full donor hematopoiesis with this treatment regimen in these patients. III. Determine the toxicity and incidence of aplasia and graft versus host disease in these patients treated with this regimen. IV. Determine the antitumor potential of this treatment regimen in these patients. V. Determine the role of NFkB in the modulation of the cytokine secretion profile of T lymphocytes during an alloimmune response in these patients treated with this regimen.

OUTLINE: Patients receive immunosuppressive medications consisting of oral mycophenolate mofetil and tacrolimus twice a day beginning on day -8 and continuing through day 45 (in the absence of graft versus host disease). Patients also receive daclizumab IV over 30 minutes on days -1, 3, and 8. Patients undergo allogeneic peripheral blood stem cell (PBSC) transplantation with donor CD34+ cells IV on day 0. If there is 0-80% donor hematopoiesis, patients receive donor lymphocyte infusions with CD3+ cells IV on days 75, 165, and 270.

PROJECTED ACCRUAL: A total of 10-45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of any of the following hematologic malignancies: Multiple myeloma Non-Hodgkin's lymphoma Indolent OR Relapsed or primary refractory high grade or intermediate grade in complete remission (CR) or partial remission (PR) after salvage chemotherapy or autologous bone marrow transplantation Hodgkin's disease Relapsed or primary refractory in CR or PR after salvage chemotherapy or autologous bone marrow transplantation Chronic lymphocytic leukemia Chronic myeloid leukemia Myelodysplastic syndrome Acute myeloid leukemia with high risk CR1 or second or greater CR Acute lymphocytic leukemia with high risk CR1 or second or greater CR Must have a 6 antigen HLA identical sibling donor Must have one of the following conditions that confer an increased risk for undergoing allogeneic bone marrow transplantation after myeloablative preparative regimen: Over 55 years of age AST or ALT greater than 2.5 times upper limit of normal (ULN) Bilirubin greater than 1.8 times ULN Renal dysfunction with creatinine greater than 1.5 mg/dL (after 12 courses of prior cytotoxic therapy) Undergone one or more prior autologous bone marrow transplantations Refuse to undergo allogeneic bone marrow transplantation using a myeloablative preparative regimen A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: See Disease Characteristics Renal: See Disease Characteristics Other: Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01 (Actual); Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bijoyesh Mookerjee, MD, Study Chair — Jefferson Medical College of Thomas Jefferson University
Locations (1):
- Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland, United States